CLINICAL TRIAL: NCT03352596
Title: Effects of Low Fructose Diet on Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Low Fructose Diet in Diabetes Type 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 93567
Record Dates: First submitted 2017-11-13; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-08

CONDITIONS: Fructose Metabolism Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Eight weeks of low fructose diet with a maximum of 12 g of fructose
  Interventions: Other: low frutose diet
- control group (No Intervention): Eight weeks of regular diabetic diet with a 15%pro 30%fat 55%CHO

INTERVENTIONS:
Other: low frutose diet
  Arms: intervention group

SUMMARY:
Diabetes is one of the most common and chronic diseases in the world, with the prevalence and incidence of this disease rising in most societies, especially in Iran. Suitable treatments for type 2 diabetes include changing lifestyle with exercise, nutrition, and drug use. New research suggests that added sugar, especially fructose, is the main trigger for diabetes and pre-diabetes even more potent than other carbohydrates. Fructose has a low glycemic index (23μg =) and slowly increases blood glucose levels. Therefore, it is thought that replacing fructose instead of glucose can have a positive effect on glycemic control of diabetic patients..

ELIGIBILITY:
Inclusion Criteria:

1. Age of 70-40 years
2. body mass index(BMI) between 18.5 and 27
3. Type 2 diabetes People who only control their diabetes by using glucose lowering tablets Type 2 diabetes (1 to 10 years)

Exclusion Criteria:

1. Pregnancy and lactation
2. Thyroid gland disorders
3. Kidney disease and inflammation
4. Follow the weight loss regimen 6 months before starting the study
5. Usage of fatty and fatty foods, fiber powder Vitamin A Mineral Supplements, Omega 3
6. Taking glucocorticoid drugs and non-steroidal anti-inflammatory drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
fasting blood suger(FBS) | 8 weeks
Homeostatic model assessment and insulin resistance(HOMA-IR) | 8weeks
insulin | 8 weeks

SECONDARY OUTCOMES:
Triglyceride | 8 weeks
Total cholestrole | 8 weeks
LDL-C | 8 weeks
HDL-C | 8 weeks
Blood pressure | 8 weeks